CLINICAL TRIAL: NCT06315335
Title: A SINGLE CENTER, RANDOMIZED, INVESTIGATOR- AND PARTICIPANT-BLIND, PLACEBO-CONTROLLED, PARALLEL-GROUP, ETHNOBRIDGING PHASE 1 STUDY TO EVALUATE SAFETY, TOLERABILITY, AND PHARMACOKINETICS AFTER SINGLE-DOSE OF UCB9741 IN HEALTHY CAUCASIAN AND JAPANESE PARTICIPANTS
Brief Title: A Study to Assess the Safety and Pharmacokinetics of a Single Dose of UCB9741 in Healthy Caucasian and Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UP0118
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants
Keywords: Phase 1; UCB9741

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort 1 (Caucasian) (Experimental): Study participants enrolled in this arm will receive either injections (sc) of the lowest dose level of UCB9741 or Placebo
  Interventions: Drug: UCB9741; Drug: Placebo
- Cohort 2 (Japanese) (Experimental): Study participants enrolled in this arm will receive either subcutaneous (sc) injections of the lowest dose level of UCB9741 or Placebo
  Interventions: Drug: UCB9741; Drug: Placebo
- Cohort 3 (Caucasian) (Experimental): Study participants enrolled in this arm will receive either subcutaneous (sc) injections of the highest dose level of UCB9741 or Placebo
  Interventions: Drug: UCB9741; Drug: Placebo
- Cohort 4 (Japanese) (Experimental): Study participants enrolled in this arm will receive either subcutaneous (sc) injections of the highest dose level of UCB9741 or Placebo
  Interventions: Drug: UCB9741; Drug: Placebo
- Cohort 5 (Caucasian) (Experimental): Study participants enrolled in this arm will receive either subcutaneous (sc) injections of the highest dose level of UCB9741 (using a different volume per injection than cohort 3) or Placebo
  Interventions: Drug: UCB9741; Drug: Placebo

INTERVENTIONS:
Drug: UCB9741 — Pharmaceutical form: Solution Participants will receive UCB9741 during the Treatment Period.
Drug: Placebo — Pharmaceutical form: Solution Participants will receive Placebo during the Treatment Period.

SUMMARY:
The purpose of the study is investigate the safety, tolerability and pharmacokinetic of UCB9741 after 2 dose strengths administered subcutaneous as a single-dose in healthy Caucasian and Japanese participants.

ELIGIBILITY:
Inclusion criteria:

For all subjects:

* Male or female between 18 to 55 years old, overtly healthy
* Female participants must not be pregnant or breastfeeding
* Female participants must be either of non-childbearing potential or using a highly efficient birth control method
* Male participants must use acceptable contraception and refrain from sperm donation during the study 90 days
* Body mass Index within the range 18 to 30 kg/m^2 (inclusive)

For Japanese subjects only:

Japanese descent as evidenced in appearance and verbal confirmation of familial heritage and is of Japanese descent with all 4 grandparents

For Caucasian subjects only:

Caucasian descent as evidenced in appearance and verbal confirmation of familial heritage and is of Caucasian descent with all 4 grandparents

Exclusion criteria:

* Participant has a known hypersensitivity to any components of the investigational medicinal product (IMP) or other biologic drugs or humanized antibodies (mAbs)
* Participant has clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe posttreatment hypersensitivity reactions
* Participant has abnormal blood pressure (BP) (outside the normal range)
* Participant has alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) >1.5x upper limit of normal (ULN)
* Participant has a recent history or currently active clinically-significant bacterial, fungal, endoparasite, or viral (including hospitalization for coronavirus disease 2019 (COVID-19)) infection (within 6 months of the Screening Visit)
* Participant has a history of inflammatory bowel disease (includes Crohn's disease and ulcerative colitis)
* Participant has a history of diabetes
* Study participant has a corrected QT interval (QTc) >450msec for male study participants or >470msec for female study participants
* Participant has sensitivity to heparin or heparin-induced thrombocytopenia
* Participant has a positive test for substance of abuse, or is a regular alcohol consumer defined as an average weekly intake of >14 units
* Participant has received any prescription or nonprescription medicines within 14 days (or 5 half-lives of the respective drug, whichever is longer) prior to the Baseline Visit, other than contraceptives or occasional use of analgesic
* Participant has received Bacillus Calmette-Guerin vaccinations within 1 year prior to the Baseline Visit or within 90 days after the final dose of investigational medicinal product (IMP)
* Participant has been treated with biologic agents (such as mAbs, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to the Baseline Visit
* Participant has participated in another study of an IMP within the previous 90 days or 5 half-lives of the IMP (whichever longer), or is currently participating in another study of an IMP

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of TEAEs | From Baseline Visit up to the End of Study Visit (Week 8)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. Treatment emergent adverse events (TEAEs) are adverse events not present prior to the pharamceutical product administration or an already present event that worsens either in intensity or frequency
Occurrence of treatment-emergent SAEs | From Baseline up to the End of Study Visit (Week 8)
  A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  Results in death Is life-threatening Requires inpatient hospitalisation or prolongation of existing hospitalisation Results in persistent or significant disability/incapacity, or Is a congenital anomaly/birth defect Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above

SECONDARY OUTCOMES:
Cmax | From Day 1 (predose) up to the End of Study Visit (Week 8)
  Cmax: Maximum serum concentration
AUC0-t | From Day 1 (predose) up to the End of Study Visit (Week 8)
  AUC0-t: Area under the curve from 0 to the time of the last quantifiable concentration
AUCinf | From Day 1 (predose) up to the End of Study Visit (Week 8)
  AUCinf: Area under the curve from 0 to infinity

CONTACTS AND LOCATIONS:
Locations (1):
- Up0118 10001, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.